CLINICAL TRIAL: NCT04296526
Title: Barriers to Participation in Physical Activity Among University Students: Which Intervention? Two-phase Study Using Transteoretic Model
Brief Title: Two-phase Transteoretic Model Research for Participation in Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Saliha Gürdal Karakelle, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 99984023-302.20.03
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Sedentary Behavior
Keywords: physical activity; transtheoretical model; university students
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Precontemplation (Experimental)
  Interventions: Behavioral: Exercise Prescription; Behavioral: Exercise Education; Behavioral: Social Support
- Contemplation (Experimental)
  Interventions: Behavioral: Exercise Prescription; Behavioral: Exercise Education; Behavioral: Social Support
- Preparation (Experimental)
  Interventions: Behavioral: Exercise Prescription; Behavioral: Exercise Education; Behavioral: Social Support

INTERVENTIONS:
Behavioral: Exercise Prescription — To prescribe exercise programs that can be easily applied at home/dormitory/living place for students.
  Other Names: Social Support
Behavioral: Exercise Education — To organize sessions for how to proper exercise.
Behavioral: Social Support — Supports such as peer influence or reminder phone messages

SUMMARY:
The purpose of the first phase of this study is to determine the physical activity (PA) barriers and motivational factors of university students and their body awareness using the transteoretic model (TTM).

The aim of the second phase of the study is to evaluate the effectiveness of interventions aimed at eliminating barriers determined in students who are in the "precontemplation", "contemplation" and "preparation" stages according to TTM. Also it will be examined the effects of these interventions on PA level.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being educated at the Faculty of Health Sciences
* Being volunteer

Exclusion Criteria:

* Being audial and vision impaired
* Having orthopedic, neurological and metabolic problems that will prevent physical activity
* Being unable to communicate in Turkish
* No pedometer program on the smartphone or using it for less than 1 year

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Exercise: Stages of Change (Short Form) | Change from baseline at 8 weeks.
  It consists of the question "Do you exercise regularly?" and five answers. These answers are "precontamplation", "contemplation", "preparation", "action" and "maintanence".

SECONDARY OUTCOMES:
Exercise Barrier Scale | At baseline and 8th weeks
  It was developed in response to a need for an instrument to determine perceptions of individuals concerning the barriers to participating in exercise.
International Physical Activity Questionnaire - Short Form | At baseline and 8th weeks
  IPAQ-SF provides information on walking, moderate and vigorous activities and time spent sitting, within a week.
Motivation Scale For Participation In Physical Activity | At baseline and 8th weeks
  It is a measurement tool to measure the motivation of students to participate in physical activity.
Body Awareness Questionnaire | At baseline and 8th weeks
  he BAQ is an 18-item scale designed to assess self-reported attentiveness to normal nonemotive body processes, specifically, sensitivity to body cycles and rhythms, ability to detect small changes in normal functioning, and ability to anticipate bodily reactions.
Number of steps in weekly | At baseline and 1-2-3-4-5-6-7-8th weeks
  Number of steps in weekly will be recorded by smartphone application.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No